CLINICAL TRIAL: NCT03054922
Title: Impact of Intraoperative Fluid Management on Electrolyte and Acid-base Variables
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, David P. Martin, Director, Acute Pain Services, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-01093
Record Dates: First submitted 2017-02-13; First posted 2017-02-16 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline (Active Comparator): 0.9% Sodium Chloride
  Interventions: Drug: Normal Saline
- Lactated Ringers (Active Comparator): Each 100 mL of Lactated Ringer's Injection USP contains:
  Sodium Chloride USP 0.6 g; Sodium Lactate USP 0.31 g; Potassium Chloride USP 0.03 g; Calcium Chloride Dihydrate USP 0.02 g; Water for Injection USP qs
  Interventions: Drug: Lactated Ringer
- Normosol-R (Active Comparator): Each 100 mL of Normosol-R contains sodium chloride, 526 mg; sodium acetate, 222 mg; sodium gluconate, 502 mg; potassium chloride, 37 mg; magnesium chloride hexahydrate, 30 mg.
  Interventions: Drug: Normosol-R Inj

INTERVENTIONS:
Drug: Normal Saline — IV infusion of 0.9% NaCl throughout surgery.
  Other Names: 0.9% NaCl
  Arms: Normal Saline
Drug: Lactated Ringer — IV infusion of lactated ringer throughout surgery.
  Arms: Lactated Ringers
Drug: Normosol-R Inj — IV infusion of Normosol throughout surgery.
  Arms: Normosol-R

SUMMARY:
During major surgical procedures, intravascular volume is maintained with the administration of isotonic fluids such as Lactated Ringers (LR), Normal Saline (NS) or Normosol-R. All three of these fluids are in common clinical use for this purpose. As large volumes of NS may result in a dilutional acidosis and an increasing base deficit, it may cloud clinical decision making when resuscitative efforts are guided by acid-base status on routine arterial blood gas analysis. This is a prospective, randomized study to evaluate changes in acid-base and electrolyte (sodium, potassium, calcium) status with the use of various isotonic fluids for intraoperative resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Major surgical procedure requiring arterial access

Exclusion Criteria:

* Comorbid disease process that contraindicates the use of any 1 of the 3 crystalloid solutions.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactated Ringers: Each 100 mL of Lactated Ringer's Injection USP contains:
  Sodium Chloride USP 0.6 g; Sodium Lactate USP 0.31 g; Potassium Chloride USP 0.03 g; Calcium Chloride Dihydrate USP 0.02 g; Water for Injection USP qs
  Lactated Ringer: IV infusion of lactated ringer throughout surgery.
Period: Overall Study
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Started | 20 | 19 | 20
Completed | 20 | 19 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (3) | 14 (2) | 14 (2) | 14 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 14 | 41
  Male | 3 | 9 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59
Weight [Mean (Standard Deviation); unit: kilograms] | 61 (13) | 57 (19) | 57 (18) | 58 (17)

OUTCOME MEASURES:

1. Primary Outcome: Change in Base Deficit
Description: Change in base deficit from 1st to 2nd blood gas to measure metabolic acidosis
Time Frame: During surgery (typically 4-6 hrs in length)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Number analyzed (Participants) | 20 | 19 | 20
mEq/L | -1.5 (2.4) | -1.2 (2.3) | -0.5 (1.5)

2. Secondary Outcome: Change in Sodium
Description: Change in sodium electrolyte from 1st to 2nd blood gas
Time Frame: During surgery (typically 4-6 hrs in length)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Number analyzed (Participants) | 20 | 19 | 20
mEq/L | 0.1 (1.7) | -0.4 (1.5) | -0.1 (1.9)

3. Secondary Outcome: Change in Potassium
Description: Change in potassium electrolyte from 1st to 2nd blood gas
Time Frame: During surgery (typically 4-6 hrs in length)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Number analyzed (Participants) | 20 | 19 | 20
mEq/L | 0.4 (0.4) | 0.7 (0.6) | 0.2 (0.4)

4. Secondary Outcome: Change in Ionized Calcium
Description: Change in calcium electrolyte from 1st to 2nd blood gas
Time Frame: During surgery (typically 4-6 hrs in length)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Number analyzed (Participants) | 20 | 19 | 20
mEq/L | 0.01 (0.05) | -0.13 (0.57) | -0.01 (0.08)

5. Secondary Outcome: Change in pH
Description: Change in pH from 1st to 2nd blood gas
Time Frame: During surgery (typically 4-6 hrs in length)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
Number analyzed (Participants) | 20 | 19 | 20
units on a scale | -0.03 (0.04) | -0.02 (0.06) | 0.01 (0.06)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Normal Saline | Lactated Ringers | Normosol-R
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT03054922/Prot_SAP_000.pdf